CLINICAL TRIAL: NCT02741739
Title: A Randomized, Open-Label, Parallel Group Study of the Pharmacokinetics, Safety, and Tolerability of a Single Subcutaneous Dose of REGN1033 Produced From Two Different Cell Lines in Healthy Subjects
Brief Title: Study of the Blood Concentrations of Two Formulations of REGN1033 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R1033-HV-1503
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Drug concentration; REGN1033; blood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference Drug (Experimental): REGN1033 Reference Formulation
  Interventions: Drug: REGN1033
- Test Drug (Experimental): REGN1033 Test Formulation
  Interventions: Drug: REGN1033

INTERVENTIONS:
Drug: REGN1033

SUMMARY:
Primary Objective: Determine blood concentrations of two formulations of REGN1033.

Secondary Objective: Assess safety and tolerability of REGN1033.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy males and females (not of childbearing potential) between the ages of 18 and 65 years
2. Body weight between 50.0 kg and 95.0 kg
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide signed informed consent

Key Exclusion Criteria:

1. Donation or loss of approximately 400 mL or more of blood within 8 weeks prior to dosing, or plasma up to 14 days prior to dosing
2. Hemoglobin not within normal limits
3. Positive drug and alcohol screen test results at screening visits 1 and 2
4. Low or elevated blood pressure and/or heart rate after 3 minutes resting in the seated position:
5. Recent use (within 3 months prior to screening) of androgenic steroids
6. Participation in any clinical research study that evaluated another investigational drug or therapy within 30 days or at least 5 half-lives, whichever is longer, of the investigational drug, prior to the screening visit
7. Previous exposure to any biological therapeutic agent, except vaccines
8. Known sensitivity to tamoxifen, doxycycline, or similar compounds (ie, tetracyclines)
9. Pregnant or breastfeeding women, and women of childbearing potential
10. Sexually active men who are unwilling to practice adequate contraception during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Serum REGN1033 concentration-time curve (AUC) | Pre-dose to day 57
Peak REGN1033 concentration (Cmax) | Pre-dose to day 57

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) from baseline to the end of the study | Day 1 to end of study (Day 57)
Presence or absence of anti-drug antibody (ADA) | Day 1 to end of study (Day 57)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- San Antonio, Texas, United States